CLINICAL TRIAL: NCT00686790
Title: An Open Label, Uncontrolled, Study to Assess the Response of Peg-Intron in naïve Patients With Chronic Hepatitis B and D Co-infection
Brief Title: Efficacy of Peginterferon Alfa-2b in Previously Untreated Subjects With Chronic Hepatitis B and D Co-infection (Study P04603)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04603
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2011-01-17 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis D, Chronic; Hepatitis B, Chronic
Keywords: Hepatitis D; Hepatitis B
MeSH Terms: conditions — Hepatitis D, Chronic; Hepatitis B, Chronic; Hepatitis D; Hepatitis B | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PegIntron (Experimental): All participants received PegIntron (Peginterferon alfa-2b) weekly based on their body weight.
  Interventions: Biological: Peginterferon alfa-2b (PegIntron, SCH 54031)

INTERVENTIONS:
Biological: Peginterferon alfa-2b (PegIntron, SCH 54031) — Peginterferon alfa-2b 1.5 mcg/kg/wk subcutaneously (SC) for 52 weeks.
  Other Names: SCH 54031, PegIntron

SUMMARY:
The objective of this study is to determine the effectiveness of peginterferon alfa-2b 1.5 mcg/kg/week administered for 52 weeks (wk) in previously untreated participants coinfected with hepatitis virus B and D. After 52-week treatment and 52-week follow-up, the virologic, biochemical, and histological response will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Participants must demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent.
* Age 18-65 years old.
* HBsAg positive >6 months.
* ALT >= 2 ULN >6 months.
* HDV RNA positive serology.
* Serum antibody to hepatitis delta antigen of IgG and IgM class.
* Knodell score HAI >= 6 and F >= 0; positive test for intrahepatic Delta antigen in liver biopsy.
* Women of childbearing potential (includes women who are less than 1 year postmenopausal and women who become sexually active) must be using an acceptable method of birth control (e.g., hormonal contraceptive, medically prescribed IUD, condom in combination with spermicide) or be surgically sterilized (e.g., hysterectomy or tubal ligation).
* Participants must be free of any clinically significant disease (other than chronic hepatitis B and D), that would interfere with study evaluations.
* Participants must understand and be able to adhere to the dosing and visit schedules, and agree to record symptom severity scores, medication times, concomitant medications, and adverse events accurately and consistently in a daily diary.

Exclusion Criteria:

* Age <18 and >65.
* Concomitant HCV and/or HIV infection.
* Actual liver failure (total serum bilirubin >2.5 x normal, prolonged prothrombin time >3 sec, serum albumin <3 g/dl, history of ascites, variceal bleeding, or hepatic encephalopathy).
* Toxic or autoimmune hepatitis (ANA titers > 1:160), metabolic liver diseases (Wilson disease, hemochromatosis, α-1 antitrypsin deficiency)
* Women who are pregnant or nursing.
* Leukopenia (<2500/mm^3), neutropenia (<1000/mm^3), hemoglobin <10 g/dl, presence of other severe diseases (myocardiopathy, diabetes mellitus, arterial hypertension, neoplasia, neurologic diseases, malnutrition).
* Antiviral, immunomodulatory, corticosteroid, or chemotherapeutical treatment within 6 months of the participation in the study.
* Depression and/or psychiatric disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2005-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the enrolled participants, 19 received no study medication and 1 was not eligible. The Intent-to-Treat (ITT) population is 48.
Groups:
- PegIntron: Peginterferon alfa-2b 1.5 mcg/kg/wk SC for 52 weeks
Period: Overall Study
Arm/Group | PegIntron
Started | 48
Completed | 32
Not Completed | 16
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1
Not completed — Lost to Follow-up | 12

BASELINE CHARACTERISTICS:
Arm/Group | PegIntron
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: years] — ITT Population
  years | 37.55 (12.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 26
Region of Enrollment [Number; unit: Participants]
  Romania | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Virological Response
Description: For virological response, a participant was defined as a responder if his/her serum sample tested negative for Hepatitis D Virus - ribonucleic acid (HDV-RNA) by polymerase chain reaction (PCR) at end of treatment (EOT).
Time Frame: 52 weeks (end of treatment [EOT]), 104 weeks (end of follow-up [EOF]) following treatment initiation
Population: The population analyzed excludes participants that were not administered any study medication and had protocol violations. 2 participants with adverse events (AE) that had protocol violations have been included in the analysis.
Measure: Number; unit: Participants
Arm/Group | PegIntron
Number analyzed (Participants) | 36
Participants
  Responders at 52 weeks | 12
  Non-responders at 52 weeks | 24
  Responders at 104 weeks | 9
  Non-responders at 104 weeks | 27

2. Secondary Outcome: Number of Participants With Hepatitis B Virus (HBV) Replication Response (HBV Response)
Description: Serum samples collected from the participants were tested by PCR to detect HBV-DNA. HBV response was defined as the absence of HBV-deoxyribonucleic acid (HBV-DNA) in serum.
Time Frame: 52 week (EOT)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | PegIntron
Number analyzed (Participants) | 36
Participants
  Responders | 6
  Non responders | 30

3. Primary Outcome: Number of Participants With a Biochemical Response
Description: A participant was defined as a responder if his alanine aminotransferase (ALT) level after 52 weeks, i.e. at EOT, was below the upper reference range as specified by Bioclinica. The normal reference range for ALT is 5-55 U/L.
Time Frame: 52 weeks (EOT), 104 weeks (EOF)
Population: The population analyzed excluded participants that were not administered study medication, had protocol violations and those for whom ALT values were not available.
  2 participants with adverse events (AE) that had protocol violations have been included in the analysis.
Measure: Number; unit: Participants
Arm/Group | PegIntron
Number analyzed (Participants) | 32
Participants
  Responders at 52 weeks | 18
  Non-responders at 52 weeks | 14
  Responders at 104 weeks | 9
  Non-responders at 104 weeks | 23

4. Primary Outcome: Number of Participants With a Combined Response
Description: The combined response was defined as an ALT level below the upper
  reference range and a negative HDV-RNA test. The normal reference range for ALT is 5-55 U/L.
Time Frame: 52 weeks (EOT), 104 weeks (EOF)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | PegIntron
Number analyzed (Participants) | 32
Participants
  Responders at 52 weeks | 7
  Non-responders at 52 weeks | 25
  Responders at 104 weeks | 6
  Non-responders at 104 weeks | 26

5. Secondary Outcome: Number of Participants With a Liver Histology Response
Description: The liver histology response was defined as at least a 2 point decrease in the necrosis inflammation score (a sum of periportal necrosis [0-10], lobular inflammation [0-4], portal inflammation [0-4], with the total score of 18 representing the worst outcome) and no increase or regression of fibrosis (scored [0-4]) in the pre- and post-treatment liver biopsies.
  The efficacy of treatment based on histological response was assessed by the investigator as complete response, partial response, minimal response, progressive disease, and not assessable at EOT.
Time Frame: Baseline and 52 week (EOT)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | PegIntron
Number analyzed (Participants) | 36
Participants
  Complete response | 10
  Partial response | 14
  Minimal response | 6
  Progressive disease | 3
  Response not assessable | 3

ADVERSE EVENTS:
Description: Adverse events are reported for all 48 participants that received study medication and included the ITT population, as well as one participant that was identified to be ineligible for the study after enrollment.
Arm/Group | PegIntron
Serious Adverse Events (participants affected / at risk) | 3/49
Other Adverse Events (participants affected / at risk) | 47/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegIntron (N=49)
PANCREATITIS (Gastrointestinal disorders) | 1 (1)
PYREXIA (General disorders) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegIntron (N=49)
VERTIGO (Ear and labyrinth disorders) | 9 (86)
VISION BLURRED (Eye disorders) | 3 (15)
ABDOMINAL PAIN (Gastrointestinal disorders) | 9 (32)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 (3)
DIARRHOEA (Gastrointestinal disorders) | 5 (7)
DRY MOUTH (Gastrointestinal disorders) | 3 (11)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 4 (8)
NAUSEA (Gastrointestinal disorders) | 18 (94)
VOMITING (Gastrointestinal disorders) | 7 (20)
ASTHENIA (General disorders) | 16 (76)
CHEST PAIN (General disorders) | 4 (13)
CHILLS (General disorders) | 32 (187)
FATIGUE (General disorders) | 26 (135)
INFLUENZA LIKE ILLNESS (General disorders) | 4 (21)
IRRITABILITY (General disorders) | 7 (24)
PYREXIA (General disorders) | 38 (310)
ANOREXIA (Metabolism and nutrition disorders) | 14 (43)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 22 (231)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 (4)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 5 (56)
MYALGIA (Musculoskeletal and connective tissue disorders) | 32 (253)
DIZZINESS (Nervous system disorders) | 15 (94)
HEADACHE (Nervous system disorders) | 38 (674)
SOMNOLENCE (Nervous system disorders) | 5 (26)
ANGER (Psychiatric disorders) | 5 (15)
DEPRESSION (Psychiatric disorders) | 3 (5)
INSOMNIA (Psychiatric disorders) | 6 (10)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 (3)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 6 (21)
ALOPECIA (Skin and subcutaneous tissue disorders) | 8 (15)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 3 (7)
PRURITUS (Skin and subcutaneous tissue disorders) | 4 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review.